CLINICAL TRIAL: NCT01844726
Title: Functional Neuroimaging Effects of the N-methyl-D-aspartate Receptor (NMDAR) Partial Agonist, GLYX-13, on Learning and Memory in Healthy Individuals
Brief Title: Effects of GLYX-13 on Learning and Memory in Healthy Individuals and Those With Psychiatric Illness
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study sponsor was acquired by another company.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, James Reilly, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU77430
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Psychiatric Illness; Healthy
Keywords: healthy individuals; schizophrenia; schizoaffective disorder; learning; memory; cognitive enhancement; fMRI
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Psychotic Disorders | interventions — GLYX-13 peptide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLYX-13 (Experimental): Single IV infusion of GLYX-13, 5mg/kg,
  Interventions: Drug: GLYX-13
- Placebo (Placebo Comparator): Single IV administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLYX-13 — Single injection (5 mg/kg) of GLYX-13, an NMDAR partial agonist
  Arms: GLYX-13
Drug: Placebo — Single injection of placebo (saline)
  Arms: Placebo

SUMMARY:
The present study proposes to evaluate the potential cognitive enhancing effects of GLYX-13, an NMDAR partial agonist, among a group of healthy adults and those with psychiatric illness on a series of functional magnetic resonance imaging (fMRI) learning and memory tasks.

DETAILED DESCRIPTION:
In a single blind randomized parallel group design, we will evaluate the whether a single dose of GLYX-13 vs. placebo increases cognitive performance on tasks of learning, declarative memory, and working memory, and associated task-related increases in blood oxygen level-dependent (BOLD) activation in hippocampus and dorsolateral prefrontal cortex, respectively. Positive findings will provide biomarker evidence for GLYX-13 effects on neural systems underlying these cognitive processes.

ELIGIBILITY:
Inclusion Criteria:

For all Individuals

* Male and female subjects
* Ages 18 - 40 years
* General intellectual abilities falling broadly within the average range (estimated intelligence quotient (IQ) between 80 - 119)
* Sufficient ability to understand study requirements and provide written informed consent

For Patients

-Diagnosis of Schizophrenia or Schizoaffective Disorder

Exclusion Criteria:

For all individuals:

* History of neurologic disorder or systemic medical condition that may interfere with central nervous system function
* History of seizures
* History of heard injury with loss of consciousness or concussion
* Positive screen for drugs of abuse: cocaine, marijuana, phencyclidine, ketamine, opioid, or other agent that is being abused in the opinion of the investigator
* Females who are currently pregnant or plan to become pregnant during the study period
* History of allergy, sensitivity, or intolerance to N-methyl-D-Aspartate receptor (NMDAR) ligands including ketamine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone
* History of any ferromagnetic object in the body
* Presence of any medical device or implant for which MRI is contraindicated including cardiac pacemaker, aneurysm clip, cochlear implant, copper intrauterine device (IUD), neurostimulator, or any other device deemed unsafe
* Bullet or shrapnel in body
* Metallic braces or permanent retainer
* Significant claustrophobia

For Healthy Individuals

* Personal history of any Axis I disorder according to the Structured Clinical Interview for the DSM-5 (SCID-5) criteria
* History of treatment with antidepressant, antipsychotic, stimulant,sedative/ hypnotic, mood stabilizing, or anticholinergic medications or lithium
* History among first-degree family members of any psychotic illness or major mood disorder (e.g., major depressive disorder, recurrent; bipolar I or II disorder)

For Patients

* Treatment with Clozaril
* Change in medication within 1 month
* Hospitalization within 1 month

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Reilly, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GLYX-13 | Placebo
Started | 22 | 22
Completed | 21 | 21
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Excessive motion in MRI resulted in discontinuation. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLYX-13 | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (4.5) | 25.2 (5.0) | 26.2 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42
Estimated Intelligence Quotient (IQ) [Mean (Standard Deviation); unit: units on a scale] — Estimated Intelligence Quotient (IQ) reflects the standardized reading score from the Wide Range Achievement Test - 4th version (WRAT4), which is commonly used as a proxy for estimated IQ. This score has a population mean of 100 and standard deviation (SD) of 15, with higher scores reflective of higher estimated IQ. In the current protocol, subjects had estimated IQ scores falling broadly within the average range ((minimum) 80 - (maximum)119).
  units on a scale | 105.7 (9.2) | 107.9 (8.8) | 106.8 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Change in fMRI BOLD Signal During a Category Learning Task
Description: Evidence of enhanced functional magnetic resonance imaging (fMRI) blood oxygen level-dependent (BOLD) signal change during a category learning task among individuals receiving GLYX-13 administration compared to those receiving placebo.
  Value represents fMRI BOLD signal change (in % change) across a task derived functional network. Higher scores indicate greater task-based activation across this functional circuit.
Time Frame: within 1 hour of administration
Measure: Mean (Standard Deviation); unit: percentage of BOLD signal change
Arm/Group | GLYX-13 | Placebo
Number analyzed (Participants) | 21 | 21
percentage of BOLD signal change | .16 (.16) | .08 (.15)
Statistical Analysis 1: Comparison: GLYX-13 vs Placebo; Change in BOLD signal activation across task derived learning circuit were compared between GLYX-13 and placebo groups using an independent group t-test; Test type: Superiority; p = .10, t-test, 2 sided; Mean Difference (Net) = .05

2. Secondary Outcome: Category Learning Behavioral Performance
Description: This measure reflects the percentage of correct trials on a category learning task in which subjects learned the category membership (group A or group B) of 8 three-digit numbers presented over 64 trials. Higher values (>50%) reflect increased accuracy in learning the category membership.
Time Frame: within 1 hour of administration
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Arm/Group | GLYX-13 | Placebo
Number analyzed (Participants) | 21 | 21
percentage of correct trials | 72.5 (16.4) | 75.2 (14.0)
Statistical Analysis 1: Comparison: GLYX-13 vs Placebo; Test type: Superiority; p = .57, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | GLYX-13 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 9/21 | 9/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLYX-13 (N=21) | Placebo (N=21)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (Nervous system disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Palpitation (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection discomfort (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No